CLINICAL TRIAL: NCT03204773
Title: Studying Non-motor Symptoms in Patients With Hereditary Spastic Paraplegia (HSP) Compared to Healthy Controls
Brief Title: Studying Non-motor Symptoms in HSP
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Tim W. Rattay, Assistant doctor and postdoctoral researcher, University Hospital Tuebingen
Other Study IDs: NMS in HSP
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: SPG4

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HSP patients: Patients with hereditary spastic paraplegia regardless of their genetic mutation
  Interventions: Diagnostic Test: EuroQol five dimensions questionaire (EQ-5D); Diagnostic Test: Modified Fatigue Impact Scale (MFI); Diagnostic Test: Brief Pain Inventory (BPI); Diagnostic Test: Becks Depression Inventory (BDI); Diagnostic Test: Restless-leg Questionaire (RLS diagnostic criteria)
- Healthy controls: healthy controls (spouses, relatives, or other healthy controls)
  Interventions: Diagnostic Test: EuroQol five dimensions questionaire (EQ-5D); Diagnostic Test: Modified Fatigue Impact Scale (MFI); Diagnostic Test: Brief Pain Inventory (BPI); Diagnostic Test: Becks Depression Inventory (BDI); Diagnostic Test: Restless-leg Questionaire (RLS diagnostic criteria)

INTERVENTIONS:
Diagnostic Test: EuroQol five dimensions questionaire (EQ-5D) — Testing quality of life.
Diagnostic Test: Modified Fatigue Impact Scale (MFI) — Screening for fatigue
Diagnostic Test: Brief Pain Inventory (BPI) — Testing for pain
Diagnostic Test: Becks Depression Inventory (BDI) — Screening for depression
Diagnostic Test: Restless-leg Questionaire (RLS diagnostic criteria) — Testing for restless-legs

SUMMARY:
Comparing the non-motor symptoms of patients with hereditary spastic paraplegia (HSP) to healthy controls (spouses, relatives or other healthy controls) by using the a number of specific questionaires

DETAILED DESCRIPTION:
https://lamapoll.de/NMS_in_HSP

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Patients with HSP (hereditary spastic paraplegia)
* Group 2: Healthy controls
* Age 18 to 70 years
* Written, informed consent

Exclusion Criteria:

* Lack of ability for a written, informed consent
* Presence of spastic gait disorder or other neurological condition (Group 2)

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We recruit known patients to our department or via patient interest groups.
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Identification of relevant non-motor symptoms in SPG4 | day 1
  By using the five mentioned scales we try to identify relevant non-motor symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Tim W. Rattay, MD, Principal Investigator — Researcher
Locations (1):
- University Hospital Tübingen, Center for Neurology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rattay TW, Boldt A, Volker M, Wiethoff S, Hengel H, Schule R, Schols L. Non-motor symptoms are relevant and possibly treatable in hereditary spastic paraplegia type 4 (SPG4). J Neurol. 2020 Feb;267(2):369-379. doi: 10.1007/s00415-019-09573-w. Epub 2019 Oct 23. PMID 31646384
- See also: Link Citation (DOI) — https://doi.org/10.1007/s00415-019-09573-w